CLINICAL TRIAL: NCT06676553
Title: INtraprocedural Feedback-Optimized Renal Denervation Based on Measurements Obtained Through Renal Artery Stimulation: a Randomized Controlled Proof-of-concept Trial to Assess Whether Renal Denervation Guided by Renal Artery Stimulation Outperforms Conventional Renal Denervation in 6-month Ambulatory Blood Pressure Reductions
Brief Title: INtraprocedural Feedback-Optimized Renal Denervation Based on Measurements Obtained Through Renal Artery Stimulation: a Randomized Controlled Trial (INFORM)
Acronym: INFORM
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Smart Health Technology Research and Development Center, National Taiwan University (Unknown); Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202405100RIPE; ERP-2023-13518 (Other Grant/Funding Number: Medtronic)
Record Dates: First submitted 2024-11-04; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Hypertension, Uncontrolled; Hypertension, Resistant; Hypertension
Keywords: Hypertension; Renal denervation; Electric stimulation; Renal artery; Radiofrequency ablation
MeSH Terms: conditions — Hypertension | interventions — Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- A: Renal artery stimulation-induced systolic blood pressure rise suppressed (<20 mmHg) (No Intervention): No further renal denervation after standard renal denervation procedure
- B: Re-denervation if renal artery stimulation-induced systolic blood pressure rise not suppressed (Active Comparator): Another round of renal denervation (main renal artery for positive proximal stimulation; branch artery for positive distal stimulation) after standard renal denervation. The definition of non-suppressed is systolic blood pressure rise >=20 mmHg compared to baseline.
  Interventions: Device: Radiofrequency ablation alone, re-denervation to main and/or branch renal artery
- C: Control if renal artery stimulation-induced systolic blood pressure rise not suppressed (Placebo Comparator): No further renal denervation after standard renal denervation. The definition of non-suppressed is systolic blood pressure rise >=20 mmHg compared to baseline.
  Interventions: Procedure: Radiofrequency ablation alone, no further renal denervation

INTERVENTIONS:
Device: Radiofrequency ablation alone, re-denervation to main and/or branch renal artery — Re-denervation according to the site where renal artery stimulation can induce systolic blood pressure rise of >= 20 mmHg. Main renal artery denervation if proximal main renal artery stimulation positive, while branch renal artery denervation if distal main renal artery stimulation positive.
  Arms: B: Re-denervation if renal artery stimulation-induced systolic blood pressure rise not suppressed
Procedure: Radiofrequency ablation alone, no further renal denervation — No further renal denervation after standard renal denervation even renal artery stimulation-induced systolic blood pressure rise >= 20 mmHg
  Arms: C: Control if renal artery stimulation-induced systolic blood pressure rise not suppressed

SUMMARY:
Our previous study (Huang HC, Pan HY, Wang TD, Circ Cardiovasc Interv 2023;16:e012779) demonstrated that when renal artery stimulation continues to trigger systolic blood pressure increases (>=20 mmHg increase compared to baseline) after the initial procedure, patients show poor blood pressure reduction 6 months following renal denervation. Based on this finding, we designed a proof-of-concept trial comparing two approaches: a guided strategy versus conventional renal denervation. In the guided strategy, we perform additional ablations of main and/or branch renal arteries if immediate post-procedure stimulation still elevates systolic blood pressure (>=20 mmHg increase compared to baseline). The conventional approach involves no repeat procedures. This trial aims to determine whether the guided strategy leads to better clinical outcomes, measured by 6-month ambulatory blood pressure changes, and to establish the value of using intraprocedural feedback to assess and guide renal denervation treatment.

DETAILED DESCRIPTION:
1. Anesthesia: Intravenous propofol to achieve adequate sedation throughout the course.
2. Renal artery stimulation (RAS) will be performed at 2 sites (proximal and distal main renal artery) in both renal arteries. Pacing frequency was set at 10 Hz, pacing output at 20 mA with a pulse duration of 10 ms, and duration of 60 sec based on earlier researches. The maximal systolic blood pressure rise and branch renal artery constriction since the start of RAS till 3 minutes after its discontinuation will be recorded. The body reaction during RAS will be recorded (0, no response; 1, mild (voice) response; 2. limited movement; 3. significant movement).
3. Renal denervation (RDN) will be performed using the multielectrode Symplicity Spyral RDN catheter. The multielectrode RDN catheter contains 4 electrodes separated from each other in a spiral configuration. Up to 4 discrete radiofrequency (RF) ablations were applied simultaneously. Each application lasts ≤60 s with a power ≤8 Watts (W) and a target temperature of ≤70°C (158°F). Electrodes that do not reach the therapeutic temperature or impedance drop are automatically switched off.
4. Post RDN renal artery stimulation:

After RDN completed, renal artery stimulation will be repeated immediately. The maximal RAS-induced SBP changes will be recorded. All BP readings are the average of 8 consecutive beats by default (Siemens, Germany), which could minimize the inadvertent BP fluctuations by movements and respiration (8 beats could encompass at least one respiratory cycle). The branch renal artery constriction since the start of RAS till 3 minutes after its discontinuation will be recorded. The body reaction during RAS will be recorded (0, no response; 1, mild (voice) response; 2. limited movement; 3. significant movement).

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypertension and are willing to undergo renal denervation.
* Patients are treated with antihypertensive medications, or with an office systolic blood pressure (SBP) >140 mm Hg or diastolic blood pressure (DBP) >90 mm Hg, and 24-hour SBP of >130 mmHg or DBP >80 mm Hg, irrespective of antihypertensive treatment.

Exclusion Criteria:

* An unsuitable renal artery anatomy for renal denervation, assessed by computed tomographic angiography (main renal artery lumen diameter <3 mm or a total length <20 mm).
* Secondary hypertension, including hyperaldosteronism, pheochromocytoma, and renal artery stenosis (>50% stenosis in one or both arteries).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
24-hour systolic blood pressure reduction (compared to baseline) | 6 months following the index renal denervation

SECONDARY OUTCOMES:
24-hour diastolic blood pressure reduction (compared to baseline) | 6 months following the index renal denervation
Awake and asleep systolic/diastolic blood pressure and heart rate changes (compared to baseline) | 6 months following the index renal denervation
Serum creatinine and estimated glomerular filtration rate changes | 6 months following the index renal denervation

OTHER OUTCOMES:
24-hour blood pressure changes based on branch artery constriction following renal artery stimulation | 6 months following the index renal denervation
24-hour blood pressure reduction (compared to baseline) | 1 year and 2 years following the index renal denervation

CONTACTS AND LOCATIONS:
Overall Officials: Tzung-Dau Wang, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Under reasonable request and approved by the principle investigator, the information could be shared.
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Result] Huang HC, Pan HY, Wang TD. Renal Nerve Stimulation Predicted Blood Pressure-Lowering Responses to Percutaneous Renal Denervation. Circ Cardiovasc Interv. 2023 Feb;16(2):e012779. doi: 10.1161/CIRCINTERVENTIONS.122.012779. Epub 2023 Feb 21. No abstract available. PMID 36802802